CLINICAL TRIAL: NCT01404416
Title: Effect of Antenatal Iron-contained Multiple Micronutrient Supplementation, Cesarean Delivery, and CDMR on Child Health- A Post-trial Follow-up Chinese Study
Brief Title: Effect of Antenatal Iron-contained Multiple Micronutrient Supplementation, Cesarean Delivery, and CDMR on Child Health
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Liu Jianmeng, Institute of Reproductive and Child Health, Peking University
Other Study IDs: 5119001
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Overweight/Obesity; Anemia; Mental Development
MeSH Terms: conditions — Overweight; Obesity; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The follow-up study was based on our previous nutritional intervention trial entitled "Impact of Prenatal Vitamin/Mineral Supplements on Perinatal Mortality (NCT00133744)". We followed up all livebirths born to women of the trial to measure their height, weight, and hemoglobin and to implement a questionaire survey (including developmental milestones, disease history, breast feeding, passive smoking, et al). We selected a sub-sample of infants to assess their IQ, emotional and behavioral problem, and language development status. The outcomes of interest include death, body mass index, overweight/ obesity, stunting/ wasting/ thinness, anemia, developmental milestones, IQ, emotional and behavioral disorder, language developmental status, and disease history. Other interesting exposure includes breast feeding, passive smoking, et al. We hypothesize that intrauterine nutritional exposure has an impact on offspring's physical, mental, and language development. We also hypothesize that cesarean delivery including CDMR has an impact on offspring's these outcomes.

DETAILED DESCRIPTION:
The follow-up study was based on our previous nutritional intervention trial entitled "Impact of Prenatal Vitamin/Mineral Supplements on Perinatal Mortality (NCT00133744)". We followed up all livebirths born to women of the trial to measure their height, weight, and hemoglobin and to implement a questionaire survey (including developmental milestones, disease history, breast feeding, passive smoking, et al). We selected 1200 <30 months infants to assess their IQ with Bayley scale, emotional and behavioral problem with CBCL scale, and language development status with LDS scale. We also selected 1500 >30 months children to measure their emotional and behavioral problem with CBCL scale. The exposure groups include intrauterine nutritional exposure and cesarean delivery exposure as well as CDMR. The outcomes of interest include death, body mass index, overweight/ obesity, stunting/ wasting/ thinness, anemia, developmental milestones, IQ, emotional and behavioral disorder, language developmental status, and disease history. Other interesting exposure includes breast feeding, passive smoking, et al. We hypothesize that intrauterine nutritional exposure has an impact on offspring's physical, mental, and language development. We also hypothesize that cesarean delivery including CDMR has an impact on offspring's these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all livebirths

Exclusion Criteria:

* died
* moved out
* refused to participate
* being incapable of participation

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all livebirths born to women of our previous trial (NCT00133744) who were from Laoting, Fengrun, Xianghe, Mancheng, and Yuanshi counties of China.
Sampling Method: Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Mancheng Maternal and Child Health Hospital, Baoding, Hebei
  - Xianghe Maternal and Child Health Hospital, Langfang, Hebei
  - Yuanshi Maternal and Child Health Hospital, Shijiazhuang, Hebei
  - Fengrun Maternal and Child Health Hospital, Tangshan, Hebei
  - Laoting Maternal and Child Health Hospital, Tangshan, Hebei

REFERENCES:
- [Derived] Si KY, Li HT, Zhou YB, Li ZW, Zhang L, Zhang YL, Ye RW, Liu JM. Cesarean delivery on maternal request and common child health outcomes: A prospective cohort study in China. J Glob Health. 2022 Feb 26;12:11001. doi: 10.7189/jogh.12.11001. eCollection 2022. PMID 35265334